CLINICAL TRIAL: NCT03648580
Title: Intervention for the Elderly With Malnutrition, Hidden Hunger and Low Skeletal Muscle Mass in Binhu Community Hospital of Nanjing
Brief Title: Intervention for the Elderly With Malnutrition, Hidden Hunger and Low Skeletal Muscle Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Ting Zhao, Technologist-in-charge, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JYX201603
Record Dates: First submitted 2017-12-20; First posted 2018-08-27 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Malnutrition Risk in Elder

STUDY DESIGN:
Intervention Model Description: the subjects will be randomized into intervention group and control group.
Masking Description: It's an open study. The number of protocol evaluable subjects for each group that complete the study and comply well with study protocol is planned to be 30.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Give the verbal nutrition education and supply Ensure Complete powder that will be the oral nutrition supplement, with the dose of 6 scoops (53.8 grams) twice daily.Duration: 12 weeks
  Interventions: Dietary Supplement: Ensure Complete powder; Other: verbal nutrition education
- Control group (Other): just give the verbal nutrition education.
  Interventions: Other: verbal nutrition education

INTERVENTIONS:
Dietary Supplement: Ensure Complete powder — Supply the Ensure Complete powder that will be the oral nutrition supplement, with the dose of 6 scoops (53.8 grams) twice daily.Duration: 12 weeks
  Arms: Intervention group
Other: verbal nutrition education — give the verbal nutrition education

SUMMARY:
Background: As the aging of the population aggravating, the ratio of the elderly in empty nest family has reached 50%, particularly in big and medium size cities, it is as high as 70%. The elderly in those families where no child living inside, elderly living alone, including an individual living alone or living with spouse are known as empty nester. The diversity of food consumption of empty nester is always poor, with single and simple meals, especially for the consumption of "core food" (fish, meat, egg, milk, vegetables and fruits), and the quantity and variety of consumption is very limited, which make the elderly be prone to be deficient of high quality protein and micronutrient. In 2005, the World Health Organization (WHO) brought up a new concept for the universally exiting problem of vitamin and trace elements intake deficiency among people, namely Hidden Hunger. With age increasing, multiple causes such as single eating pattern, empty nest lifestyle and chronic diseases lead to long term intake deficiency of protein and micronutrient of the elderly, which will further result in various symptoms of nutritional deficiency. Therefore, it is particularly important for the empty nester to have sufficient energy, high quality protein and multiple micronutrients to prevent hidden hunger and sarcopenia, thus avoiding the health problem and life quality decreasing caused by them.

ELIGIBILITY:
Inclusion Criteria:

1. the one who is or is between 65 to 85 years old, male or female;
2. the one with nutritional risk according to MNA-Short Form evaluation (score less than12);
3. the one who has low skeletal muscle mass (with bioelectrical impedance analysis report indicating that the skeletal muscle mass is less than 90% of the normal level) and/or the one who has at least 1 type of the micronutrient deficiency symptom (part A < 40 or part A < 85 in the hidden hungry evaluation questionnaire)

Exclusion Criteria:

1. long-term bedridden or the one has difficult in taking food orally;
2. Liver failure in recent one year;
3. Renal insufficiency (serum creatinine is more than 2 times of normal value)
4. the one who is allergic to or not applicable to the component in oral dietary supplement;
5. the one with parkinsonism, epilepsy and other nervous system disorders;
6. malignant tumor patients with chemotherapy and chemotherapy;
7. irritable bowel disease and other chronic wasting diseases.
8. Taking multi-vitamin&mineral supplements or protein or other oral nutritional supplements

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Mini Nutritional Assessment short-form (MNA®-SF) score | 12 weeks
  MNA®-SF is a validated nutrition screening and assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition. The Screening score(max. 14 points) is 12-14 points indicates "Normal nutritional status", 8-11 points indicates "At risk of malnutrition", 0-7 points indicates "Malnourished".

SECONDARY OUTCOMES:
Muscle mass--The change of percentage of skeletal muscle mass | 12 weeks
  The skeletal muscle mass of the participants were assessed using a multiple-frequency bioelectrical impedance analysis (BIA) instrument (InBodyS10; InBody, Shanghai, China). Percentage of skeletal muscle mass (PSM) is the ratio of skeletal muscle mass to ideal skeletal muscle mass which is defined according to the height and the standard BMI of each patient. Normal PSM standard is defined as values in the range of 90-110%. We defined low skeletal muscle mass (Sarcopenia) as values <90% of the standard.
The change of BMI | 12 weeks
  Weight in kilograms was measured during the study. Height in meters was measured at the baseline. Weight and height will be combined to report BMI in kg/m^2.
Muscle strength--The change of Calf circumference | 12 weeks
  Calf circumference(CCF) was measured with a soft tape, the measurement standard is divided into less than 31 cm and 31 cm or greater.
Muscle strength--The change of Grip strength | 12 weeks
  Grip strength with a calibrated grip force meter to measure the grip strength of the dominant hand. The cut-off of grip strength is 26 kg for men and 18 kg for women.
Muscle strength--6 meters gait speed | 12 weeks
  A standard stopwatch is used to measure the subject's 6 meters gait speed for 3 times, and the average pace is then calculated. The intercept value of step speed is 0.8m/s.
Hidden Hunger Assessment Scale | 12 weeks
  There are two parts in Hidden Hunger Assessment Scale. Part A includes the options for 10 dietary behaviors, giving 3 behavioral frequency choices (> 3 times per week, 5 points; 1 to 3 times per week, 3 points; never, 0 points), score ranges from 0 to 50 which are evaluated and classified into three categories. Part B includes 17 options on the manifestation of micronutrient deficiencies, giving three frequencies of occurrence to score (consecutive, 0 points; occasionally, 3 points; never, 5 points). The result ranges from 0 to 85, while different ranges were evaluated and defined differently. The scores of Part A and B of the participants were summed up and separated into three definition: <70 as "obvious hunger requesting immediate intervention", 70-123 as "existing hidden hunger requesting improvement", and > 123 as "no hidden hunger ".
Dietary Nutrients | 12 weeks
  Average daily intake of dietary nutrients
The change of DETERMINE score | 12 weeks
  The DETERMINE is checklist to find out if someone you know is at nutritional risk. The checklist is based on warning signs described. DETERMINE is the first letter of all warning signs: Disease, Eating poorly, Tooth loss/month pain, Economic hardship, Reduced social contact, Multiple medicines, Involuntary weight loss/gain, Needs assistance in self care, Elder years above age 80.
  The total score is 21. 0-2 scores means good, recheck your nutritional scores in 6 months.
  3-5 scores you are at moderate nutrition risk. Recheck your nutritional scores in 3 months.
  6 or more scores means you are at high nutrition risk. Bring this checklist the next time you see your doctor, dietitian or other qualified health or social service professional. Talk with them about any problem you may have. Ask for help to improve your nutritional health.
Questionnaire--Healthy lifestyle questionnaire | 12 weeks
  Healthy lifestyle questionnaire be designed by investigator. 24 questions cover healthy lifestyle, that are about disease, fallen, infection, allergy, drink alcohol, smoke, eating habit, activity intensity/frequency, sleep quality, emotion etc.
Questionnaire--Self-satisfaction questionnaire | 12 weeks
  The self-satisfaction questionnaire be completed by subject. The questionnaires be used to evaluate self-rate satisfaction for stool pattern, sleep, health status, quality of life, energy level, vitality level, daily activities. There are some questions to get the state of the stool pattern and sleep. Others are evaluated in the percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Zhao, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China